CLINICAL TRIAL: NCT00456820
Title: Wellbutrin XL Effects on SSRIs Induced Changes in the Reactivity of the Frontal Cortex and Limbic System to Emotional Stimuli: An fMRI Study
Brief Title: Wellbutrin XL Effects on SSRIs Induced Changes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0406-27; 45-870-26
Record Dates: First submitted 2005-09-14; First posted 2007-04-05 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-04

CONDITIONS: Depression; Side Effects; Sexual Dysfunction; Apathy
Keywords: Mood Regulating Circuit; SSRI; fMRI
MeSH Terms: conditions — Depression; Sexual Dysfunction, Physiological; Lethargy | interventions — Bupropion

INTERVENTIONS:
Drug: Wellbutrin XL

SUMMARY:
The purpose of this study is to find out differences in activation of mood regulating areas of the brain in response to negative and positive pictures, before and after 6 weeks of additional Wellbutrin XL treatment. Participants should have been treated for depression with an SSRI medication (e.g., Prozac, Zoloft, Paxil, Celexa or Lexapro) and have decreased depression symptoms but also be experiencing side effects of medications such as sexual side effects and feelings of apathy (indifference, lack of interest) and lack of full emotional response. We will first take a brain scan to measure activity in different parts of the brain, while subjects are seeing pictures, using Magnetic Resonance Imaging (MRI) scan. Then we will add Wellbutrin XL - another well-known antidepressant that acts by increasing the chemical dopamine in the brain, to subjects' treatment. Wellbutrin addition is useful in decreasing the sexual side effects of SSRIs. After treatment with Wellbutrin XL for 6 weeks subjects will have a second MRI scan with picture rating.

DETAILED DESCRIPTION:
Hypotheses:

Hypothesis 1.After wellbutrin XL addition for 6 weeks, SSRI treated subjects will show increased activation and connectivity of prefrontal cortex and limbic regions such as the amygdala on exposure to negative and positive pictures

Hypothesis 2.Increase in activation of the MRC (Mood Regulating Circuit) will correlate with decrease in Apathy Evaluation Scale (AES) score and Sexual Dysfunction Score.

We plan to study a maximum of 15 subjects in this study. SSRI treated depressed patients who after treatment of depression continue to suffer from sexual dysfunction and apathy will be included in the study. fMRI will be conducted at baseline and after addition of Wellbutrin XL treatment 300 mg po qd and then used at a dose of 300 mg - 450 mg from week 3 - 6 depending on response and tolerance. Patients will also be rated weekly on 17-item Hamilton Depression Rating Scale, Montgomery-Asberg Depression Rating Scale (MADRAS) (Montgomery and Asberg 1979), AES (Marin et al 1991), Changes in Sexual Functioning Questionnaire (CSFQ) and Clinical Global Impression (Improvement) weekly for 6 weeks. Depressed patients will also be rated on the scan days on cognitive measures such as verbal memory and working memory.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 - 60 years and able to give voluntary informed consent.
2. Satisfy criteria for recent treatment with for Major Depressive Episode using DSM-IV episode recently treated with an adequate dose of an SSRI (sertraline, paroxetine, fluoxetine, citalopram, escitalopram) with 17-item Hamilton Depression Rating Scale (HDRS) score < 18.
3. Complaining of symptoms of apathy, lack of feeling or sexual dysfunction with AES score < 10 and/or MADRAS item 8 (inability to feel > 1) and/or CSFQ score > 10
4. Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire. 5) Able to be managed as outpatients for initial assessment and during treatment as ascertained by the following - Symptoms not worsening by more than 10 points on the HDRS during the course of the study and not representing danger to self or others.

Exclusion Criteria:

1. Meeting DSM-IV criteria for bipolar disorder, schizophrenia, schizophreniform disorder, schizoaffective disorder, atypical psychosis, primary anxiety disorder, mental retardation, or organic mental (including organic mood) disorder.
2. Use of neuroleptic in the past 1 year.
3. History of seizure disorder
4. History of eating disorders such as bulimia or anorexia nervosa
5. History of lack of response or intolerance to bupropion.
6. Use of mood stabilizers in the past 2 weeks.
7. Use of benzodiazepines in the past 2 weeks.
8. Acutely suicidal or homicidal or requiring inpatient treatment.
9. Meeting DSM-IV criteria for other substance dependence, including alcohol within the 6 months, except caffeine or nicotine. The criteria will be evaluated by interview and urinary toxicology screening initially and on test days.
10. Use of alcohol in the past 1 week.
11. No serious medical or neurological illness as assessed by physical examination and laboratory examination including CBC and blood chemistry.
12. Abnormal TSH values. If on synthroid should be on a stable dose for 3 months prior to the study with no changes during the study.
13. Current pregnancy or breast-feeding.
14. Metallic implants.
15. Previously known positive HIV blood test (as latent central dysfunction may be present) as reported by the subject.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15
Dates: Start 2004-07; Study Completion 2007-11

PRIMARY OUTCOMES:
Activation and connectivity of frontal cortex and limbic region as measured by MRI scan at baseline and six weeks from baseline
Improvement of scores on Apathy Evaluation Scale and Changes in Sexual Functioning Questionnaire given weekly for six weeks

SECONDARY OUTCOMES:
Improvement of scores on Hamilton Depression Rating Scale given weekly for six weeks
Improvement on Clinical Global Impression Severity and Improvement Scales given weekly for six weeks
Improvement of scores on MADRS (specifically item #8) given weekly for six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Adult Psychiatry Clinic, Indianapolis, Indiana, United States